CLINICAL TRIAL: NCT01337362
Title: Recurrent Hypoglycaemia in Type 1 Diabetes: Effects on Cognitive Function, Cerebral Electrical Activity, and Skin Temperature
Brief Title: Recurrent Hypoglycaemia in Type 1 Diabetes
Acronym: HypoNeuro
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hillerod Hospital, Denmark (Other)
Collaborators: University of Southern Denmark (Other); Rigshospitalet, Denmark (Other); UNEEG Medical A/S (Industry)
Responsible Party: Principal Investigator, Anne-Sophie Sejling, MD, Hillerod Hospital, Denmark
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: H-1-2011-024
Record Dates: First submitted 2011-03-30; First posted 2011-04-18 (Estimated); Last update posted 2014-10-16 (Estimated); Status verified 2014-10

CONDITIONS: Hypoglycaemia
Keywords: Diabetes; Hypoglycaemia; EEG; Thermography; Hypoglycaemia-associated autonomic failure; QTc interval; Hypoglycemic alarm device; Hormone response
MeSH Terms: conditions — Hypoglycemia; Diabetes Mellitus | interventions — Insulin; Constriction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Patients with hypoglycemia awareness (Active Comparator): Patients who have symptoms when the blood sugar level is low
  Interventions: Procedure: Insulin clamp
- patients with hypoglycaemic unawareness. (Experimental): Patients who do not feel any symptoms when the blood sugar levels are low
  Interventions: Procedure: Insulin clamp

INTERVENTIONS:
Procedure: Insulin clamp — Patients will be exposed to low bloodsugar
  Other Names: Insulin; clamp

SUMMARY:
Patients with type 1 diabetes are at risk of very low blood sugar levels (hypoglycaemia) as a severe side effect to insulin therapy, in particular subjects who have lost warning of hypoglycaemia. During hypoglycaemia a low frequent activity can be seen with electroencephalography (EEG) as cognitive function declines.

The purpose of the study is to investigate the activity in the brain, the cognitive function, and the skin temperature when patients are exposed to repeated hypoglycaemia. The results will show whether the response to hypoglycaemia will change after repeated episodes.

It is our hope that results can contribute to improved understanding of hypoglycaemic EEG changes.

DETAILED DESCRIPTION:
Background:

Patients with type 1 diabetes are at risk of severe hypoglycaemia as a severe side effect to insulin therapy, in particular subjects who have lost warning of hypoglycaemia (hypoglycaemia unawareness). The episodes are associated with impaired quality of life and can lead to permanent brain damage and death.

During hypoglycaemia a low frequent activity can be seen with electroencephalography (EEG) as cognitive function declines. Repeated hypoglycaemic episodes result in down regulation of counter regulatory and symptomatic responses. It is not known whether a similar phenomenon is present for cerebral dysfunction as judged by EEG changes and cognitive function.

The purpose is to investigate the activity in the brain, the cognitive function, and the skin temperature when patients are exposed to repeated hypoglycaemia. The results will show whether the response to hypoglycaemia will change after repeated episodes.

The methods:

The investigators will recruit two groups of patients: Patients with hypoglycemia awareness and patients with hypoglycaemic unawareness.

The patients are exposed to hypoglycaemia on two concomitant days while the investigators record EEG and perform cognitive tests. Skin temperature is assessed by the use of thermography. If the patient has hypoglycaemic unawareness a 4 week period follows where the glycaemic control is loosened to avoid hypoglycaemia episodes and the patients is then exposed to hypoglycaemia again.

The prospect:

It is the investigators hope that results can contribute to improved understanding of hypoglycaemic EEG changes and skin temperature changes. This could be of potential benefit for patients with hypoglycaemic unawareness.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes
* Age > 18 years
* - Have had diabetes for more than 5 years
* Negative pregnancy test
* Caucasian
* Signed written informed consent

Exclusion Criteria:

* Pregnant or breastfeeding
* Epilepsy
* Self-perceived impaired hearing
* Use of antiepileptic medicine
* Use of neuroleptics within the last 6 months
* Use of benzodiazepines within the last month
* Use of betablockers
* Previous stroke or other disease in the brain
* Cardiovascular disease
* Alcohol-, drug- or medicine abuse
* Previous allergic reaction to heparin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2011-05; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
EEG | 2 years
  EEG will be analysed in order to see whether there are any differences between aware and unaware patients during hypoglycaemia. It is our hope that the result can help develop an alarm before the patient experiences severe hypoglycaemia.

SECONDARY OUTCOMES:
QTc interval | 2 years
  The investigators want to investigate whether the QTc complex gets wider during hypoglycaemia. This is in order to see whether long QTc could be the explanation behind sudden dearth in diabetes patients.
Skin temperature | 2 years
  Skin temperature will be measured by thermography. The investigators want to see whether the skin can be used as a biomarker for hypoglycaemia.
Auditory evoked potentials | 2 years
  The investigators what to see whether there is any difference in auditory evoked potentials (AEP) between aware and unaware diabetic patients. The subject will hear a common and a rare sound in a 4:1 ratio while the EEG is recorded. Afterwards the data is analyzed and the AEPs are addressed.
Cognitive function | 2 years
  The investigators want to address whether there are any differences in the cognitive function between aware and unaware patients. The cognitive function will be addressed by the use of cognitive function tests (CalCAP) and Stroops tests as well.

CONTACTS AND LOCATIONS:
Overall Officials: Anne-Sophie Sejling, MD, Principal Investigator — Hillerod Hospital
Locations (1):
- Hillerod Hospital, Hillerød, Hillerød, Denmark

REFERENCES:
- [Derived] She R, Al-Sari NH, Mattila IM, Sejling AS, Pedersen J, Legido-Quigley C, Pedersen-Bjergaard U. Decreased branched-chain amino acids and elevated fatty acids during antecedent hypoglycemia in type 1 diabetes. BMJ Open Diabetes Res Care. 2023 Jun;11(3):e003327. doi: 10.1136/bmjdrc-2023-003327. PMID 37369531
- [Derived] Rubega M, Sparacino G, Sejling AS, Juhl CB, Cobelli C. Hypoglycemia-Induced Decrease of EEG Coherence in Patients with Type 1 Diabetes. Diabetes Technol Ther. 2016 Mar;18(3):178-84. doi: 10.1089/dia.2015.0347. Epub 2016 Jan 8. PMID 26745007